CLINICAL TRIAL: NCT00595504
Title: Phase IV Study of Ramelteon as an Adjunct Therapy in Non-Diabetic Patients With Schizophrenia
Brief Title: Ramelteon as an Adjunct Therapy in Non-Diabetic Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, David C. Henderson, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007P-001929; FWA00003136
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
Keywords: schizophrenia; metabolism; antipsychotics; diabetes; rozerem
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Diabetes Mellitus | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ramelteon 8mg/day
  Interventions: Drug: Ramelteon
- 2 (Placebo Comparator): sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Two week supply of ramelteon 8mg/day first dispensed at baseline. New two week supply of study medication dispensed at each biweekly visit for 8 consecutive weeks.
  Other Names: Rozerem
  Arms: 1
Drug: Placebo — Two week supply of placebo tablets first dispensed at baseline. New two week supply of placebo dispensed at each biweekly visit for 8 consecutive weeks.
  Arms: 2

SUMMARY:
This study involves people who have schizophrenia or schizoaffective disorder who are currently taking antipsychotic medications. Some antipsychotic medications may cause weight gain and may increase the risk of diabetes mellitus and heart disease.The purpose of this study is to find out what happens if another medication (ramelteon) is used along with your antipsychotic medication. We want to find out whether doing this will:

* Change the way your body breaks down fat and sugar.
* Affect your waist size, stomach fat and triglycerides (a type of fat in your blood).
* Improve how your body responds to insulin.
* Affect your quality of sleep.
* Reduce movement disturbances Ramelteon is approved by the U.S. Food and Drug Administration (FDA) to treat people that have difficulty falling asleep. It is not approved for such things as affecting waist size or improving how the body breaks down fat and sugar. Its use in this study is investigational.

DETAILED DESCRIPTION:
This is an 8-week randomized, double blind, placebo-controlled pilot study with 4- week follow up assessment, of ramelteon 8 mg/day, administered to subjects for 8 consecutive weeks as an adjunctive therapy in 40 non-diabetic schizophrenia subjects to examine ramelteon effects on body composition, glucose and lipid metabolism, sleep quality and symptoms of tardive dyskinesia using the Massachusetts General Hospital General Clinical Research Center. As far as we know, no previous study has been done to explore the potential role of ramelteon in improving metabolic, sleep, and movement disturbances in schizophrenia subjects. The novel approach of adjunctive ramelteon treatment in the schizophrenia population is promising.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia, schizoaffective disorder, any subtype or schizophreniform disorder
* male or female, age 18-65 years
* treatment with clozapine, olanzapine, quetiapine or risperidone
* well established compliance with medications
* Body Mass Index (BMI) of > 27 Kg/m² with any component of metabolic syndrome or insulin resistance or a BMI of > 30 Kg/m²:

Exclusion Criteria:

* inability to provide informed consent
* substance and alcohol abuse
* significant medical illness, including congestive heart failure, severe hepatic impairment, severe Chronic Obstructive Pulmonary Disease (COPD), severe sleep apnea, severe cardiovascular disease or renal disease
* current history of diabetes mellitus or thyroid disease
* women who are pregnant, breastfeeding, or who are unwilling or unable to use an effective form of birth control during the entire study
* psychiatrically unstable, patients with major depression
* patients treated with medications known to affect glucose tolerance such as birth control pills containing norgestrel, steroids, beta blockers, anti-inflammatory drugs (including daily aspirin and ibuprofen), thiazide diuretics; and agents that induce weight loss will be excluded from the study
* treatment with fluvoxamine in the or ketoconazole past two weeks
* treatment with fluconazole (a strong CYP2C9 inhibitor).
* subjects treated with ziprasidone and aripiprazole conventional agents
* treatment with sedative-hypnotics such as barbiturates, zolpidem, eszopiclone, zaleplon. The use of stable daily doses of benzodiazepines is allowed.
* known hypersensitivity to ramelteon or any of its components

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Henderson, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ananth J, Venkatesh R, Burgoyne K, Gadasalli R, Binford R, Gunatilake S. Atypical antipsychotic induced weight gain: pathophysiology and management. Ann Clin Psychiatry. 2004 Apr-Jun;16(2):75-85. doi: 10.1080/10401230490453293. PMID 15328901
- [Background] Henderson DC. Schizophrenia and comorbid metabolic disorders. J Clin Psychiatry. 2005;66 Suppl 6:11-20. PMID 16107179
- [Background] Henderson DC. Atypical antipsychotic-induced diabetes mellitus: how strong is the evidence? CNS Drugs. 2002;16(2):77-89. doi: 10.2165/00023210-200216020-00001. PMID 11825099
- [Background] Henderson DC, Copeland PM, Borba CP, Daley TB, Nguyen DD, Cagliero E, Evins AE, Zhang H, Hayden DL, Freudenreich O, Cather C, Schoenfeld DA, Goff DC. Glucose metabolism in patients with schizophrenia treated with olanzapine or quetiapine: a frequently sampled intravenous glucose tolerance test and minimal model analysis. J Clin Psychiatry. 2006 May;67(5):789-97. doi: 10.4088/jcp.v67n0513. PMID 16841629
- [Background] Casey DE, Haupt DW, Newcomer JW, Henderson DC, Sernyak MJ, Davidson M, Lindenmayer JP, Manoukian SV, Banerji MA, Lebovitz HE, Hennekens CH. Antipsychotic-induced weight gain and metabolic abnormalities: implications for increased mortality in patients with schizophrenia. J Clin Psychiatry. 2004;65 Suppl 7:4-18; quiz 19-20. No abstract available. PMID 15151456
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Newcomer JW, Haupt DW, Fucetola R, Melson AK, Schweiger JA, Cooper BP, Selke G. Abnormalities in glucose regulation during antipsychotic treatment of schizophrenia. Arch Gen Psychiatry. 2002 Apr;59(4):337-45. doi: 10.1001/archpsyc.59.4.337. PMID 11926934
- [Background] Henderson DC, Cagliero E, Copeland PM, Borba CP, Evins AE, Hayden D, Weber MT, Anderson EJ, Allison DB, Daley TB, Schoenfeld D, Goff DC. Glucose metabolism in patients with schizophrenia treated with atypical antipsychotic agents: a frequently sampled intravenous glucose tolerance test and minimal model analysis. Arch Gen Psychiatry. 2005 Jan;62(1):19-28. doi: 10.1001/archpsyc.62.1.19. PMID 15630069
- [Background] Bonora E, Kiechl S, Willeit J, Oberhollenzer F, Egger G, Targher G, Alberiche M, Bonadonna RC, Muggeo M. Prevalence of insulin resistance in metabolic disorders: the Bruneck Study. Diabetes. 1998 Oct;47(10):1643-9. doi: 10.2337/diabetes.47.10.1643. PMID 9753305
- [Background] Kitabchi AE, Temprosa M, Knowler WC, Kahn SE, Fowler SE, Haffner SM, Andres R, Saudek C, Edelstein SL, Arakaki R, Murphy MB, Shamoon H; Diabetes Prevention Program Research Group. Role of insulin secretion and sensitivity in the evolution of type 2 diabetes in the diabetes prevention program: effects of lifestyle intervention and metformin. Diabetes. 2005 Aug;54(8):2404-14. doi: 10.2337/diabetes.54.8.2404. PMID 16046308
- [Background] Lillioja S, Mott DM, Spraul M, Ferraro R, Foley JE, Ravussin E, Knowler WC, Bennett PH, Bogardus C. Insulin resistance and insulin secretory dysfunction as precursors of non-insulin-dependent diabetes mellitus. Prospective studies of Pima Indians. N Engl J Med. 1993 Dec 30;329(27):1988-92. doi: 10.1056/NEJM199312303292703. PMID 8247074
- [Background] Semenkovich CF. Insulin resistance and atherosclerosis. J Clin Invest. 2006 Jul;116(7):1813-22. doi: 10.1172/JCI29024. PMID 16823479
- [Background] Weyer C, Tataranni PA, Bogardus C, Pratley RE. Insulin resistance and insulin secretory dysfunction are independent predictors of worsening of glucose tolerance during each stage of type 2 diabetes development. Diabetes Care. 2001 Jan;24(1):89-94. doi: 10.2337/diacare.24.1.89. PMID 11194248
- [Background] Carr DB, Utzschneider KM, Hull RL, Kodama K, Retzlaff BM, Brunzell JD, Shofer JB, Fish BE, Knopp RH, Kahn SE. Intra-abdominal fat is a major determinant of the National Cholesterol Education Program Adult Treatment Panel III criteria for the metabolic syndrome. Diabetes. 2004 Aug;53(8):2087-94. doi: 10.2337/diabetes.53.8.2087. PMID 15277390
- [Background] Hayashi T, Boyko EJ, Leonetti DL, McNeely MJ, Newell-Morris L, Kahn SE, Fujimoto WY. Visceral adiposity and the risk of impaired glucose tolerance: a prospective study among Japanese Americans. Diabetes Care. 2003 Mar;26(3):650-5. doi: 10.2337/diacare.26.3.650. PMID 12610016
- [Background] Goodpaster BH, Thaete FL, Simoneau JA, Kelley DE. Subcutaneous abdominal fat and thigh muscle composition predict insulin sensitivity independently of visceral fat. Diabetes. 1997 Oct;46(10):1579-85. doi: 10.2337/diacare.46.10.1579. PMID 9313753
- [Background] Kelley DE, Thaete FL, Troost F, Huwe T, Goodpaster BH. Subdivisions of subcutaneous abdominal adipose tissue and insulin resistance. Am J Physiol Endocrinol Metab. 2000 May;278(5):E941-8. doi: 10.1152/ajpendo.2000.278.5.E941. PMID 10780952
- [Background] Jensen MD, Haymond MW, Rizza RA, Cryer PE, Miles JM. Influence of body fat distribution on free fatty acid metabolism in obesity. J Clin Invest. 1989 Apr;83(4):1168-73. doi: 10.1172/JCI113997. PMID 2649512
- [Background] Muller N, Riedel M, Gruber R, Ackenheil M, Schwarz MJ. The immune system and schizophrenia. An integrative view. Ann N Y Acad Sci. 2000;917:456-67. doi: 10.1111/j.1749-6632.2000.tb05410.x. PMID 11268373
- [Background] Maes M, Bocchio Chiavetto L, Bignotti S, Battisa Tura GJ, Pioli R, Boin F, Kenis G, Bosmans E, de Jongh R, Altamura CA. Increased serum interleukin-8 and interleukin-10 in schizophrenic patients resistant to treatment with neuroleptics and the stimulatory effects of clozapine on serum leukemia inhibitory factor receptor. Schizophr Res. 2002 Apr 1;54(3):281-91. doi: 10.1016/s0920-9964(00)00094-3. PMID 11950553
- [Background] Sirota P, Meiman M, Herschko R, Bessler H. Effect of neuroleptic administration on serum levels of soluble IL-2 receptor-alpha and IL-1 receptor antagonist in schizophrenic patients. Psychiatry Res. 2005 Apr 15;134(2):151-9. doi: 10.1016/j.psychres.2004.04.012. PMID 15840416
- [Background] Rapaport MH, Lohr JB. Serum-soluble interleukin-2 receptors in neuroleptic-naive schizophrenic subjects and in medicated schizophrenic subjects with and without tardive dyskinesia. Acta Psychiatr Scand. 1994 Nov;90(5):311-5. doi: 10.1111/j.1600-0447.1994.tb01599.x. PMID 7872033
- [Background] Naudin J, Capo C, Giusano B, Mege JL, Azorin JM. A differential role for interleukin-6 and tumor necrosis factor-alpha in schizophrenia? Schizophr Res. 1997 Aug 29;26(2-3):227-33. doi: 10.1016/s0920-9964(97)00059-5. PMID 9323355
- [Background] Lin A, Kenis G, Bignotti S, Tura GJ, De Jong R, Bosmans E, Pioli R, Altamura C, Scharpe S, Maes M. The inflammatory response system in treatment-resistant schizophrenia: increased serum interleukin-6. Schizophr Res. 1998 Jun 22;32(1):9-15. doi: 10.1016/s0920-9964(98)00034-6. PMID 9690329
- [Background] McAllister CG, van Kammen DP, Rehn TJ, Miller AL, Gurklis J, Kelley ME, Yao J, Peters JL. Increases in CSF levels of interleukin-2 in schizophrenia: effects of recurrence of psychosis and medication status. Am J Psychiatry. 1995 Sep;152(9):1291-7. doi: 10.1176/ajp.152.9.1291. PMID 7653683
- [Background] Zhang XY, Zhou DF, Cao LY, Zhang PY, Wu GY, Shen YC. Changes in serum interleukin-2, -6, and -8 levels before and during treatment with risperidone and haloperidol: relationship to outcome in schizophrenia. J Clin Psychiatry. 2004 Jul;65(7):940-7. doi: 10.4088/jcp.v65n0710. PMID 15291683
- [Background] Muller N, Riedel M, Scheppach C, Brandstatter B, Sokullu S, Krampe K, Ulmschneider M, Engel RR, Moller HJ, Schwarz MJ. Beneficial antipsychotic effects of celecoxib add-on therapy compared to risperidone alone in schizophrenia. Am J Psychiatry. 2002 Jun;159(6):1029-34. doi: 10.1176/appi.ajp.159.6.1029. PMID 12042193
- [Background] Rapaport MH, Delrahim KK, Bresee CJ, Maddux RE, Ahmadpour O, Dolnak D. Celecoxib augmentation of continuously ill patients with schizophrenia. Biol Psychiatry. 2005 Jun 15;57(12):1594-6. doi: 10.1016/j.biopsych.2005.02.024. PMID 15953498
- [Background] Sjoholm A, Nystrom T. Inflammation and the etiology of type 2 diabetes. Diabetes Metab Res Rev. 2006 Jan-Feb;22(1):4-10. doi: 10.1002/dmrr.568. PMID 15991254
- [Background] Chandalia M, Cabo-Chan AV Jr, Devaraj S, Jialal I, Grundy SM, Abate N. Elevated plasma high-sensitivity C-reactive protein concentrations in Asian Indians living in the United States. J Clin Endocrinol Metab. 2003 Aug;88(8):3773-6. doi: 10.1210/jc.2003-030301. PMID 12915668
- [Background] Monti JM, Monti D. Sleep disturbance in schizophrenia. Int Rev Psychiatry. 2005 Aug;17(4):247-53. doi: 10.1080/09540260500104516. PMID 16194796
- [Background] Correll CU, Leucht S, Kane JM. Lower risk for tardive dyskinesia associated with second-generation antipsychotics: a systematic review of 1-year studies. Am J Psychiatry. 2004 Mar;161(3):414-25. doi: 10.1176/appi.ajp.161.3.414. PMID 14992963
- [Background] Shamir E, Barak Y, Shalman I, Laudon M, Zisapel N, Tarrasch R, Elizur A, Weizman R. Melatonin treatment for tardive dyskinesia: a double-blind, placebo-controlled, crossover study. Arch Gen Psychiatry. 2001 Nov;58(11):1049-52. doi: 10.1001/archpsyc.58.11.1049. PMID 11695951
- [Background] Abilio VC, Vera JA Jr, Ferreira LS, Duarte CR, Carvalho RC, Grassl C, Martins CR, Torres-Leite D, Bignotto M, Tufik S, Ribeiro Rde A, Frussa-Filho R. Effects of melatonin on orofacial movements in rats. Psychopharmacology (Berl). 2002 Jun;161(4):340-7. doi: 10.1007/s00213-002-1081-7. Epub 2002 Apr 26. PMID 12073160
- [Background] Nishida S. Metabolic effects of melatonin on oxidative stress and diabetes mellitus. Endocrine. 2005 Jul;27(2):131-6. doi: 10.1385/endo:27:2:131. PMID 16217126
- [Background] Wolden-Hanson T, Mitton DR, McCants RL, Yellon SM, Wilkinson CW, Matsumoto AM, Rasmussen DD. Daily melatonin administration to middle-aged male rats suppresses body weight, intraabdominal adiposity, and plasma leptin and insulin independent of food intake and total body fat. Endocrinology. 2000 Feb;141(2):487-97. doi: 10.1210/endo.141.2.7311. PMID 10650927
- [Background] Raskind MA, Burke BL, Crites NJ, Tapp AM, Rasmussen DD. Olanzapine-induced weight gain and increased visceral adiposity is blocked by melatonin replacement therapy in rats. Neuropsychopharmacology. 2007 Feb;32(2):284-8. doi: 10.1038/sj.npp.1301093. Epub 2006 May 10. PMID 16710316
- [Background] Johnson MW, Suess PE, Griffiths RR. Ramelteon: a novel hypnotic lacking abuse liability and sedative adverse effects. Arch Gen Psychiatry. 2006 Oct;63(10):1149-57. doi: 10.1001/archpsyc.63.10.1149. PMID 17015817
- [Background] Monteleone P, Natale M, La Rocca A, Maj M. Decreased nocturnal secretion of melatonin in drug-free schizophrenics: no change after subchronic treatment with antipsychotics. Neuropsychobiology. 1997;36(4):159-63. doi: 10.1159/000119377. PMID 9396013
- [Background] Robinson S, Rosca P, Durst R, Shai U, Ghinea C, Schmidt U, Nir I. Serum melatonin levels in schizophrenic and schizoaffective hospitalized patients. Acta Psychiatr Scand. 1991 Sep;84(3):221-4. doi: 10.1111/j.1600-0447.1991.tb03133.x. PMID 1950621
- [Background] Evans DR, Parikh VV, Khan MM, Coussons C, Buckley PF, Mahadik SP. Red blood cell membrane essential fatty acid metabolism in early psychotic patients following antipsychotic drug treatment. Prostaglandins Leukot Essent Fatty Acids. 2003 Dec;69(6):393-9. doi: 10.1016/j.plefa.2003.08.010. PMID 14623492
- [Background] Fan X, Pristach C, Liu EY, Freudenreich O, Henderson DC, Goff DC. Elevated serum levels of C-reactive protein are associated with more severe psychopathology in a subgroup of patients with schizophrenia. Psychiatry Res. 2007 Jan 15;149(1-3):267-71. doi: 10.1016/j.psychres.2006.07.011. Epub 2006 Nov 16. PMID 17112596
- [Background] Fan X, Anderson EJ, Copeland PM, Borba CP, Nguyen DD, Freudenreich O, Goff DC, Henderson DC. Higher fasting serum insulin is associated with increased resting energy expenditure in nondiabetic schizophrenia patients. Biol Psychiatry. 2006 Dec 15;60(12):1372-7. doi: 10.1016/j.biopsych.2006.05.006. Epub 2006 Aug 22. PMID 16920075
- [Background] Ventura J, Liberman RP, Green MF, Shaner A, Mintz J. Training and quality assurance with the Structured Clinical Interview for DSM-IV (SCID-I/P). Psychiatry Res. 1998 Jun 15;79(2):163-73. doi: 10.1016/s0165-1781(98)00038-9. PMID 9705054
- [Background] Ritz R CJ: Indirect Calorimetry. Monitoring in Respiratory Care. St Louis, MO, Mosby-Yearbook, Inc, 1993
- [Background] Schakel SF, Sievert YA, Buzzard IM. Sources of data for developing and maintaining a nutrient database. J Am Diet Assoc. 1988 Oct;88(10):1268-71. PMID 3171020
- [Background] Kelly TL, Berger N, Richardson TL. DXA body composition: theory and practice. Appl Radiat Isot. 1998 May-Jun;49(5-6):511-3. doi: 10.1016/s0969-8043(97)00226-1. PMID 9569530
- [Background] Visser M, Fuerst T, Lang T, Salamone L, Harris TB. Validity of fan-beam dual-energy X-ray absorptiometry for measuring fat-free mass and leg muscle mass. Health, Aging, and Body Composition Study--Dual-Energy X-ray Absorptiometry and Body Composition Working Group. J Appl Physiol (1985). 1999 Oct;87(4):1513-20. doi: 10.1152/jappl.1999.87.4.1513. PMID 10517786
- [Background] McNamara JR, Schaefer EJ. Automated enzymatic standardized lipid analyses for plasma and lipoprotein fractions. Clin Chim Acta. 1987 Jun 30;166(1):1-8. doi: 10.1016/0009-8981(87)90188-4. PMID 3608193
- [Background] Warnick GR, Benderson J, Albers JJ. Dextran sulfate-Mg2+ precipitation procedure for quantitation of high-density-lipoprotein cholesterol. Clin Chem. 1982 Jun;28(6):1379-88. No abstract available. PMID 7074948
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Kay SR, Opler LA, Lindenmayer JP. The Positive and Negative Syndrome Scale (PANSS): rationale and standardisation. Br J Psychiatry Suppl. 1989 Nov;(7):59-67. No abstract available. PMID 2619982
- [Background] Rey JM, Hunt GE, Johnson GF. Assessment of tardive dyskinesia in psychiatric outpatients using a standardized rating scale. Aust N Z J Psychiatry. 1981 Mar;15(1):33-7. doi: 10.3109/00048678109159407. PMID 6973337
- [Background] Haro JM, Kamath SA, Ochoa S, Novick D, Rele K, Fargas A, Rodriguez MJ, Rele R, Orta J, Kharbeng A, Araya S, Gervin M, Alonso J, Mavreas V, Lavrentzou E, Liontos N, Gregor K, Jones PB; SOHO Study Group. The Clinical Global Impression-Schizophrenia scale: a simple instrument to measure the diversity of symptoms present in schizophrenia. Acta Psychiatr Scand Suppl. 2003;(416):16-23. doi: 10.1034/j.1600-0447.107.s416.5.x. PMID 12755850
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Heinrichs DW, Hanlon TE, Carpenter WT Jr. The Quality of Life Scale: an instrument for rating the schizophrenic deficit syndrome. Schizophr Bull. 1984;10(3):388-98. doi: 10.1093/schbul/10.3.388. PMID 6474101
- [Background] Hann DM, Denniston MM, Baker F. Measurement of fatigue in cancer patients: further validation of the Fatigue Symptom Inventory. Qual Life Res. 2000;9(7):847-54. doi: 10.1023/a:1008900413113. PMID 11297027
- [Background] Endicott J, Spitzer RL, Fleiss JL, Cohen J. The global assessment scale. A procedure for measuring overall severity of psychiatric disturbance. Arch Gen Psychiatry. 1976 Jun;33(6):766-71. doi: 10.1001/archpsyc.1976.01770060086012. PMID 938196
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Hoddes E, Zarcone V, Smythe H, Phillips R, Dement WC. Quantification of sleepiness: a new approach. Psychophysiology. 1973 Jul;10(4):431-6. doi: 10.1111/j.1469-8986.1973.tb00801.x. No abstract available. PMID 4719486
- [Background] Hays RD, Martin SA, Sesti AM, Spritzer KL. Psychometric properties of the Medical Outcomes Study Sleep measure. Sleep Med. 2005 Jan;6(1):41-4. doi: 10.1016/j.sleep.2004.07.006. Epub 2004 Nov 11. PMID 15680294
- [Background] Levine S. The management of resistant depression. Acta Psychiatr Belg. 1986 Mar-Apr;86(2):141-51. PMID 3088916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Freedom Trial Clinic at the Erich Lindemann Mental Health Center and were studied at the Mallinckrodt General Clinical Research Center (GCRC) at the Massachusetts General Hospital (MGH), Boston
Pre-assignment Details: After providing written informed consent, subjects underwent a diagnostic evaluation by a research psychiatrist using the Structured Clinical Interview for DSM-IV (SCID). All subjects were screened and enrolled based on eligibility criteria. Baseline study assessments were completed prior to intervention.
Groups:
- Placebo: sugar pill
Period: Overall Study
Arm/Group | Ramelteon | Placebo
Started | 16 | 9
Completed | 14 | 6
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon | Placebo | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (7) | 56 (9) | 53 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Waist Circumference
Description: A comparison between the ramelteon group and the placebo group in change in waist circumference (measured in cm) measured at Baseline and Week 8.
Time Frame: Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Ramelteon; Placebo (Sugar Pill): A double-blind, placebo-controlled, 8-week pilot trial was conducted, adding ramelteon 8 mg/day to stable outpatients with schizophrenia.
Arm/Group | Ramelteon | Placebo (Sugar Pill)
Number analyzed (Participants) | 14 | 6
cm | 106.09 (8.8) | 108.37 (6.5)

2. Primary Outcome: Change in Insulin Resistance as Measured by the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR).
Description: A comparison between the ramelteon group and the placebo group of change in insulin resistance measured by the homeostatic model assessment of insulin resistance (HOMA-IR), assessed at Baseline and Week 8.
Time Frame: Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study.
Measure: Mean (Standard Deviation); unit: HOMA score
Arm/Group | Ramelteon | Placebo (Sugar Pill)
Number analyzed (Participants) | 14 | 6
HOMA score | 2.4 (1.51) | 2.36 (1.73)

3. Primary Outcome: Change in Abdominal Fat (DEXA).
Description: A comparison between the ramelteon group and the placebo group of change in abdominal fat measured by a DEXA scan, assessed at Baseline and Week 8.
Time Frame: Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Ramelteon | Placebo (Sugar Pill)
Number analyzed (Participants) | 14 | 6
g | 3934.86 (1151.97) | 5120.92 (1770.58)

ADVERSE EVENTS:
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 0/16 | 0/9

LIMITATIONS AND CAVEATS:
The limitations of this study include the relatively small sample size and short intervention period (8 weeks).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes